CLINICAL TRIAL: NCT03673423
Title: Interobserver Variability In The Assessment Of Vascular Invasion In Pancreatic Cancer
Brief Title: Evaluation of the Interobserver Agreement on the Resectability Status of Patients With a Pancreatic Cancer
Acronym: OBTCPAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Gianpaolo Balzano, Principal Investigator, Ospedale San Raffaele
Other Study IDs: OBTCPAN
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Resectability Status; NCCN criteria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess the degree of vascular involvement is crucial in the diagnostic and therapeutic work-up of pancreatic cancer. NCCN resectability classification is used to stratify patients (in resectable, borderline resectable and non resectable) and is based on contrast-enhanced CT scan images. Unfortunately evaluation of imaging tests may rely on some degree of subjective interpretation by observers implying a fundamental variation in patient's treatments and an irreproducibility of different center study results.

This is a multicenter diagnostic study on interobserver agreement on the resectability of pancreatic cancer based upon NCCN criteria.

The primary aim of the study will be the assessment of interobserver variability to define vascular invasion and resectability status on CT scans (according to the last version of the NCCN Classification).

One hundred and thirty eight consecutive patients, able to produce an informed consent, from 18 years of age, with a non-metastatic pancreatic adenocarcinoma assessed by a contrast-enhanced high-quality CT scan will be enrolled.

69 CT scan studies provided by the centers involved (High volume for pancreatic surgery) will be randomly selected from a pool of 138 of the patients that meet the inclusion criteria. Each study will be independently reviewed by a senior radiologist and a senior surgeon of each center, blinded to patient's clinical history and CT scan report, using NCCN definition of respectability status. A CFR will be filled during the review and send to the study coordinator. The data will be than centrally analyzed to asses interobserver agreement The enrolment phase will last 6 months and the whole study will last 8 months.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma frequently invades peripancreatic major vessels (common hepatic artery, celiac axis, superior mesenteric artery and mesenteric-portal confluence), requiring vascular resection or precluding the possibility of a radical resection. To Asses local resectability in pancreatic cancer patients is a key step to the whole process of care and it can change dramatically the outcomes. It is also extremely important in the reproducibility of different scientific studies that stratified or included patients on this feature. Resectability status classification of pancreatic adenocarcinoma, according to the definition of the National Comprehensive Cancer Network (NCCN) is widely used in current surgical and oncological practice to define the degree of vascular invasion: this classification describes three different classes of tumor depending on the local extension and vascular involvement. Resectable cancers are defined when no contact with the main vessels can be detected, whereas borderline resectable and non resectable tumors have a different extent of vascular infiltration. The recommended staging exam to define vascular involvement of pancreatic adenocarcinoma is contrast-enhanced CT scan; NCCN recommends that all patients with suspicion of pancreatic adenocarcinoma have a dedicated pancreas protocol CT scan as part of the initial assessment. From the attribution of a patient to a resectability class (resectable, borderline resectable or non resectable) derives the choice of a specific therapeutic pathway, as suggested by NCCN guidelines. International validated criteria to define local respectability are available but they can be prone to subjective interpretation. An evaluation of interobserver agreement on local resectability for pancreatic cancer in a multicenter setting is needed to understand the reliability and reproducibility of this system.

The primary aim of the study will be the assessment of interobserver variability to define vascular invasion and resectability status on CT scans (according to the last version of the NCCN Classification).One senior radiologist and one senior surgeon from different Italian high-volume Institutions will separately assess the degree of vascular invasion by pancreatic cancer and the definition of resectability status according to NCCN. 69 CT scans, randomly selected from a pool of 138 studies (provided by each center and collected by the study coordinator) of non-metastatic consecutive patients with pancreatic cancers that signed the informed consent, will be evaluated. CT scans will be provided by participating centres, that will send them to the coordinating centre until reaching the planned enrolment. The images and related DVDs will be made anonymous and identified just by serial number and initials of the patient. The CT scan reports will be collected by each centre and made available by the coordinating centre for subsequent analysis. The criteria used to define the resectability status are those developed by the NCCN and included in the latest guidelines. Observers will be blinded to the CT-scan reports, as well as to the clinical history of the patient, and to the votes of the other raters. The degree of each vessel invasion and assignment of each tumor to a category of resectability status (resectable - borderline resectable - non resectable) will be defined separately by all raters, by fulfilling a template adopted and reported in NCCN guidelines. An interrater reliability analysis using the Kappa statistic will be performed to determine consistency among observers on the respectability status. The consistency among observer will be also evaluated for each point of the criteria and section of the template to asses vascular involvement in detail.

In case of significant fair or poor agreement (K < 0.50), the participating raters (consensus group), including the study coordinator, will meet to discuss the cases that will have less than 100% agreement among all the raters. Scans will be reviewed, an open discussion ensued. Based on the discussion, the consensus group will develop proposals to address the specific areas of disagreement. The CT scans not select for the first evaluation will be than evaluated, using the proposal of the consensus group by a new set of rater (one senior radiologist and one senior surgeon from each institution involved) and the new Kappa statistic will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Non-metastatic pancreatic adenocarcinoma
* Availability of contrast enhanced CT scan with adequate quality. Section thickness must be <3 mm, according to NCCN recommendations
* Pathological confirmation of pancreatic adenocarcinoma by cytology/histology is not required at the time of enrolment, but it is needed before including the CT scan in the pool of exams to be evaluated.
* Signed informed consent

Exclusion Criteria:

* Evidence of metastatic disease
* Inadequate quality CT scan (non-respecting the NCCN recommendations)
* Absence of cytology/histology confirmation
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 138 Consecutive patients, able to produce an informed consent, from 18 years of age, with a non-metastatic pancreatic adenocarcinoma assessed by a contrast-enhanced high-quality CT scan.
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-03-05 (Estimated); Study Completion 2019-05-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of interobserver variability to define vascular invasion and resectability status on CT scans | Eight months
  The primary aim of the study will be the assessment of interobserver variability to define vascular invasion and resectability status on CT scans (according to the last version of the NCCN Classification).

SECONDARY OUTCOMES:
Identification of disagreement causes and proposal of a new classification system | One year
  In case of significant low agreement (K < 0,5), causes of disagreement will be assessed and a new classification of vascular involvement will be proposed to reduce the disagreement. The new classification will be validated on the remaining 69 CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Balzano, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No